CLINICAL TRIAL: NCT04972136
Title: A Double-Blind Randomized Controlled Trial Evaluating the Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) as Treatment for Major Depressive Disorder in Transition-Age Youth With Autism Spectrum Disorder
Brief Title: rTMS for Depression in Young Adults With Autism
Acronym: rTMS-MDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Stephanie Ameis, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 141/2019
Record Dates: First submitted 2021-05-26; First posted 2021-07-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Major Depressive Disorder
Keywords: Autism Spectrum Disorder; Major Depressive Disorder; rTMS (Repetitive Transcranial Magnetic Stimulation); MRI (Magnetic Resonance Imaging); Suicidal and Self-Injurious Behaviour; Adaptive Functioning
MeSH Terms: conditions — Autism Spectrum Disorder; Depressive Disorder, Major; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active bilateral theta burst stimulation (Active Comparator): An X100 stimulator with a B65 A/P type coil (Magventure Inc.) will be used. The coil is positioned under MRI guidance using real-time neuronavigation using Brainsight [x,y,z= -38, 44, 26(left), +38, 44, 26 (right). BL-TBS will be delivered at 90% RMT, corrected for scalp to cortex distance, to targeted left and right DLPFC sites, differing only in stimulation pattern and total number of pulses (triplet 50 Hz bursts, repeated at 200 msec (i.e., 5 Hz); right DLPFC (continuous TBS, cTBS): 120 seconds uninterrupted bursts (total of 600 pulses); left DLPFC (intermittent TBS, iTBS: 2 seconds on and 8 seconds off; 600 pulses per session; total duration of 3 min 9 seconds/hemisphere).
  Interventions: Device: Active Bilateral Theta Burst Stimulation
- Sham bilateral theta burst stimulation (Sham Comparator): An X100 stimulator with a B65 A/P type coil (Magventure Inc.) will be used with the active coil facing away from the scalp, for sham stimulation. The coil is positioned under MRI guidance using real-time neuronavigation using Brainsight [x,y,z= -38, 44, 26(left), +38, 44, 26 (right). To reproduce the nociceptive qualities of the stimulation, the B65-type stimulation coil - sham side - includes a built in electrical stimulator in the coil connector which "fires" a synchronous electrical pulse along with the TMS stimulus through electrodes mounted on the forehead or near the area of stimulation, to generate auditory and somatosensory (vibration) stimuli.
  Interventions: Device: Sham Bilateral Theta Burst Stimulation

INTERVENTIONS:
Device: Active Bilateral Theta Burst Stimulation — A total of 30 active BL-TBS sessions. Stimulation will begin with right DLPFC (cTBS) followed by left DLPFC (iTBS)
  Other Names: X100 with a B65-type coil (Magventure Inc.)
  Arms: Active bilateral theta burst stimulation
Device: Sham Bilateral Theta Burst Stimulation — A total of 30 sham BL-TBS sessions. Stimulation will begin with right DLPFC (cTBS) followed by left DLPFC (iTBS)
  Other Names: X100 with a B65-type coil (Magventure Inc.)
  Arms: Sham bilateral theta burst stimulation

SUMMARY:
The current clinical trial is focused on evaluating the efficacy of rTMS for treatment of depression in youth and young adults (hereafter called transition aged youth, TAY) with autism spectrum disorder (ASD). The motivation to undertake the current efficacy study is driven by: (1) the substantial impact of depression on TAY with ASD (based on prevalence and contribution to disability/impairment); (2) lack of evidence-based treatments for depression in autism (there are no current trials rigorously evaluating any treatment for depression, i.e., psychotherapeutic, pharmacotherapeutic, brain stimulation); (3) rTMS has demonstrated efficacy in non-autistic individuals to improve symptoms of depression and may be better tolerated in youth than medication treatment; (4) a prior pilot rTMS study focused on treatment of executive function deficits in autism indicated that high frequency rTMS delivered using a rigorous randomized control trial (RCT) protocol can be feasibly implemented in TAY with autism, is well tolerated (mild to moderate adverse effects and low drop out), and has the potential to improve symptoms of depression.

DETAILED DESCRIPTION:
The investigators will use a randomized, double-blind, sham-controlled design of bilateral theta burst stimulation (BL-TBS) to dorsolateral prefrontal cortex (DLPFC) administered 5 days per week for 6 weeks (30 sessions). The investigators will recruit n=80, 16-35 year old participants with autism that do not have co-occurring intellectual disability (ID). In the current study, the target population will be individuals with autism, without ID who have co-occurring clinically significant depression. Pre/post treatment MRI will be used to study mechanisms of treatment response. The investigators will build on their previous pilot rTMS study in autism with two key innovations. First, the investigators will use theta burst stimulation (TBS) for depression as opposed to conventional rTMS. TBS is a newer form of rTMS shown to be non-inferior to conventional rTMS for depression with a similar safety profile. Tolerance of intermittent TBS (iTBS, delivered at 100% RMT to right DLPFC in ten 9-17 year-olds with ASD) has already been shown in autism in a prior open-label study. Importantly, TBS can be delivered in a fraction of the time needed for conventional rTMS. This shorter administration time may be critical for participant retention as sensory sensitivity is a major feature of autism. A shorter administration also has important practical implications for future clinical access. The investigators will use BL-TBS based on: preliminary data of improved antidepressant efficacy with a bilateral (over unilateral) TBS approach that combines left excitatory with right inhibitory DLPFC stimulation, as well as findings that bilateral (over unilateral) rTMS may improve suicidal ideation in MDD.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* ASD diagnosis confirmed by the clinician/clinical team, and IQ> or =70
* Able to participate in the informed consent process, provide voluntary informed consent and provide a spontaneous narrative description of the key elements of the study
* Clinical stability: determined by a physician, no switch of psychotropic medications or increase in dosage in the last 30 days; no change in other therapeutic interventions in last 30 days
* BDI-II score ≥21 that is sustained over a lead-in period of two weeks
* Global Assessment of Function (GAF) scores (≤60) that is sustained over a lead-in period of two weeks AND/OR VABS-III below adequate functioning at baseline assessment.

Exclusion Criteria:

* A history of a DSM-5 substance use disorder (other than tobacco) within the past six months; or a positive baseline urine drug screen
* Significantly debilitating medical or neurologic illness, or acute or unstable medical illnesses as determined by study physician
* Metal implants or a pace-maker, claustrophobia that would preclude the MRI scan
* Actively suicidal (i.e., suicidal ideation with plan and intent) or high risk for suicide as assessed by a study psychiatrist
* History of seizures
* Taking benzodiazepines at a dose greater or equal to 2mg Lorazepam or any anticonvulsant medication
* Prior rTMS treatment
* Pregnancy

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the 17-item Hamilton Rating Scale for Depression (HRSD-17) | Baseline, end of weeks 1, 2, 3, 4, 5, and 6 of treatment, and at 1-week, 4-weeks and 12-weeks post-treatment.
  The investigators will evaluate the changes in the severity of symptoms of depression before, during, and after rTMS treatment. HRSD-17 scores range from 0 to 52, with higher scores indicating greater severity of depressive symptoms (worse outcome).

SECONDARY OUTCOMES:
Change in scores on the Beck Scale for Suicide Ideation (BSI) | Baseline, end of weeks 1, 2, 3, 4, 5, and 6 of treatment, and at 1-week, 4-weeks and 12-weeks post-treatment.
  The investigators will evaluate the changes in suicidal thinking scores before, during, and after rTMS treatment. BSI scores range from 0 to 38, with higher scores indicating greater suicidal ideation (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie H Ameis, MD, MSC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No